CLINICAL TRIAL: NCT05483452
Title: Accuracy of Coplanar Template Assisted Seed Implantation for Abdominal and Pelvic Cancer
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qiu Bin, Principal Investigator, Peking University Third Hospital
Other Study IDs: ChiECRCT20220009
Record Dates: First submitted 2022-07-18; First posted 2022-08-02 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Accuracy of Coplanar Template Assisted Seed Implantation for Abdominal and Pelvic Cancer
Keywords: Coplanar Template; Abdominal and Pelvic cancer; Seed Implantation
MeSH Terms: conditions — Pelvic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, template guidance has been applied and developed in the field of puncture related operations, such as template-assisted radioactive seed implantation. With the guidance of template, needle pathway of seed implantation, biopsy and fiducial marker implantation can be precisely planned actual operation, which is conducive to the accurate proceeding. Templates can be divided into coplanar templates and non-coplanar templates. The digital coplanar template coordinate puncture system has been developed in China and has been applied in clinical practice.

In previous studies, coplanar template assisted CT-guided radioactive seed implantation has good clinical feasibility for head and neck cancer. However, the accuracy of Coplanar Template Assisted Seed Implantation for Abdominal and Pelvic cancer are lacking in prospective studies. The study aims to prospectively observe the accuracy and safety of Coplanar Template Assisted Seed Implantation for Abdominal and Pelvic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 85
2. Single or multiple abdominal or pelvic tumors (solid, partially solid)
3. Without taking drugs affecting coagulation and/or platelet aggregation are used; If used, the drug has been discontinued for a sufficient period of time (e.g. 1 week)
4. KPS>60 points with expected survival >3 months, no serious or uncontrolled underlying diseases, clinical evaluation patients can tolerate puncture
5. Planned seed implantation with applicable puncture path
6. With informed consent.

Exclusion Criteria:

1. Poor organ function (e.g. Liver decompensation)
2. The lesion close to blood vessels and intestine, or there is portal vein hypertension and superior vena cava compression, etc., which are expected to have high risks of puncture bleeding and intestinal injury
3. Poor compliance, unable to complete coordination
4. Paticipant who is considered inappropriate or unwilling to participate in this clinical trial for other reasons.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Abdominal and Pelvic cancer who are planned to undergo Coplanar Template Assisted Seed Implantation.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Dosimetry (D90) between pre-plan and post-plan | From the starting to the ending of the seed implantation (generally within 1 week).
  Dose covering 90% of target volume between pre-plan and post-plan

SECONDARY OUTCOMES:
Success rate of seed implantation | From the starting to the ending of the seed implantation (generally within 1 day).
  Success rate of seed implantation
Adverse event | Acute adverse event is defined as 1 month after seed implantation and beyond 1 month for chronic adverse event.
  Such as pneumoperitoneum, subcutaneous emphysema, hemorrhage, infection, etc.
Operating duration | From the starting to the ending of the seed implantation (generally within 2 hours)
  Operating duration from the starting to the ending
Local progression-free survival | From date of seed implantation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Local progression-free survival:Duration of the seed implantation to local tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China